CLINICAL TRIAL: NCT07367399
Title: Acute Myocardial Infarction Clinical Intelligent Decision Support System
Acronym: AMI-CIDSS
Status: Active, not recruiting | Type: Observational
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: kebingbing253
Record Dates: First submitted 2026-01-18; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Acute Myocardial Infarction; Large Language Models; Clinical Decision Support System

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Acute Myocardial Infarction (AMI) remains the leading cause of cardiovascular mortality globally. In China, while the incidence of AMI is escalating at an annual rate of 5.2%, significant clinical challenges persist: diagnostic delays in primary care facilities exceed 40%, and the "Door-to-Balloon" (D2B) compliance rate in tertiary hospitals stagnates at a mere 65%. These figures underscore systemic deficiencies, including inefficient emergency response, regional resource disparities, and fragmented longitudinal care. Although Large Language Models (LLMs) provide a transformative technical foundation for AMI management, their clinical translation is hindered by critical bottlenecks, such as non-standardized data interfaces, limited model interpretability, inadequate hardware infrastructure at the grassroots level, and the inherent tension between data privacy and training requirements.

This research proposes a comprehensive implementation strategy for an AI-driven intelligent decision-making system for AMI. On a theoretical level, the study establishes a tripartite framework of "Technological Adaptation, Scenario Implementation, and Safeguard Mechanisms." By introducing a data governance scheme based on federated learning and multimodal fusion, and constructing a "Technical-Clinical-Economic" multidimensional evaluation model, this work bridges the theoretical divide between advanced technology and clinical practice. On a practical level, the study develops adaptive gateways and lightweight models to facilitate pervasive deployment in resource-constrained settings, optimizes the full-cycle clinical workflow to improve patient outcomes, and provides a scalable, replicable pathway for implementation.

Focusing on four core challenges-technological compatibility, clinical workflow integration, the balance between privacy and performance, and the establishment of scientific evaluation systems-this research aims to surmount existing translation barriers. It seeks to enhance the quality and efficiency of AMI care while providing a seminal reference for the clinical transformation of AI in other medical specialties.

ELIGIBILITY:
Inclusion Criteria:

1. Patients meeting the diagnostic criteria for acute myocardial infarction (AMI). Acute Myocardial Infarction (AMI) encompasses both ST-segment elevation myocardial infarction (STEMI) and non-ST-segment elevation myocardial infarction (NSTEMI).

   According to the Fourth Universal Definition of Myocardial Infarction, myocardial injury is defined as the detection of an elevated cardiac troponin (cTn) value above the 99th percentile upper reference limit (URL). The injury is considered acute if there is a rise and/or fall of cTn values.

   The clinical definition of myocardial infarction (MI) requires the presence of acute myocardial injury, confirmed by abnormal cardiac biomarkers, in the setting of evidence of acute myocardial ischemia. Clinical evidence of ischemia includes at least one of the following:

   ①Symptoms of myocardial ischemia;

   ②New ischemic ECG changes;

   ③Development of pathological Q waves;

   ④Imaging evidence of new loss of viable myocardium or new regional wall motion abnormality in a pattern consistent with an ischemic etiology;

   ⑤Identification of a coronary thrombus by angiography or autopsy.
2. Patients who have provided written informed consent.

Exclusion Criteria:

1. patients with a life expectancy < 12 months due to non-cardiac comorbidities;
2. those with severe cognitive impairment hindering assessment;
3. individuals unable to comply with the long-term follow-up protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population comprised consecutive adult patients (aged ≥ 18 years) diagnosed with acute myocardial infarction (AMI) and admitted to Beijing Anzhen Hospital. AMI was defined according to the Fourth Universal Definition of Myocardial Infarction, encompassing both ST-segment elevation myocardial infarction (STEMI) and non-ST-segment elevation myocardial infarction (NSTEMI). Inclusion required documented acute myocardial injury (rise/fall of cardiac troponin above the 99th percentile URL) alongside clinical evidence of ischemia. All participants provided written informed consent. We excluded patients with a life expectancy < 12 months due to non-cardiac comorbidities, those with severe cognitive impairment hindering assessment, and individuals unable to comply with the long-term follow-up protocol. The study was approved by the Institutional Ethics Committee and conducted in strict accordance with the Declaration of Helsinki.
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Cardiac and Cerebrovascular Events (MACCE) | 1 year
  A composite endpoint comprising cardiac death, all-cause mortality, malignant arrhythmia, non-fatal recurrent myocardial infarction (MI), non-fatal stroke, unplanned repeat revascularization, and rehospitalization for heart failure.

SECONDARY OUTCOMES:
Cardiac Death | 1 year
  Defined as death resulting from a primary cardiac cause (e.g., acute MI, sudden cardiac death, heart failure, or cardiac procedures).
All-cause Mortality | 1 year
  Defined as death due to any cause, encompassing both cardiovascular and non-cardiovascular etiologies.
Non-fatal Recurrent Myocardial Infarction (MI) | 1 year
  Defined as a new myocardial infarction occurring after the index event. This includes three distinct patterns: extension of the original infarct, infarction in a region adjacent to the initial site, or a new infarction at a site distant from the original lesion.
Non-fatal Stroke | 1 year
  Consistent with the World Health Organization (WHO) definition, stroke is defined as a focal (or global) neurological deficit caused by vascular injury persisting for more than 24 hours. This includes both ischemic and hemorrhagic stroke (intracerebral, intraventricular, and subarachnoid hemorrhage).
Unplanned Repeat Revascularization | 1 year
  Defined as any non-elective readmission for percutaneous coronary intervention (PCI) or coronary artery bypass grafting (CABG).
Rehospitalization for Heart Failure | 1 year
  A complex clinical syndrome resulting from structural and/or functional cardiac abnormalities that lead to reduced cardiac output and/or elevated intracardiac pressures at rest or during stress. Diagnosis requires inpatient treatment for typical symptoms and signs, such as dyspnea, fatigue, and fluid retention (e.g., pulmonary congestion, systemic venous congestion, or peripheral edema).
Target Lesion Revascularization (TLR) | 1 year
  Defined as repeat percutaneous intervention or bypass surgery involving the target lesion, which includes the stented segment plus the 5 mm proximal and distal margins. The necessity for revascularization is indicated by: (1) target lesion stenosis >50% in the presence of objective evidence of ischemia; or (2) target lesion stenosis >70% regardless of clinical symptoms.
Target Vessel Revascularization (TVR) | 1 year
  Defined as any repeat percutaneous intervention or bypass surgery performed on any segment of the target vessel, including the target lesion, the proximal and distal segments of the main epicardial artery, and all of its branches.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Anzhen Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided